CLINICAL TRIAL: NCT02994602
Title: An Open-Label Study of Serum Testosterone and Nestorone in Females After Secondary Exposure to Nestorone ® (NES) + Testosterone (T) Combined Gel Applied to Shoulders and Upper Arms in Males: Effect of Washing or Clothing Barrier to the Application
Brief Title: Study of Serum Testosterone and Nestorone in Females After Secondary Exposure to Nestorone ® (NES) + Testosterone (T) Combined Gel Applied to Shoulders and Upper Arms in Males
Acronym: CCN005B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kimberly Myer (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of Washington (Other); Population Council (Other)
Responsible Party: Sponsor-Investigator, Kimberly Myer, Program Director, Premier Research
Organization: Premier Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCN005B; HHSN275201200002I (Other Grant/Funding Number: NICHD Contract. This is not a grant but a contract number. There is not an option to include a contract number)
Record Dates: First submitted 2016-11-18; First posted 2016-12-16 (Estimated); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy Men; Male Contraception; Healthy Women; Product Transference
Keywords: Healthy Men; Male Contraception; Healthy Women; Transfer; Transference; Gel; Nestorone; Testosterone
MeSH Terms: interventions — ST 1435

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nestorone (NES) + testosterone (T) combined gel (Experimental): A combination gel with Nestorone® (NES) and Testosterone (T) applied transdermally. The volume of gel to be applied will be approximately 5 mL. This gel volume will contain 62.5 mg of T that will deliver approximately 6 mg T to the body per day and will also contain 8.3 mg of NES that will deliver about 0.8 mg NES to the body per day (NES 8 mg/d + T 60 mg/d (NES8/T60) gel) in 5 ml of combined gel.
  Interventions: Drug: Nestorone + Testosterone Combination Gel

INTERVENTIONS:
Drug: Nestorone + Testosterone Combination Gel — The combined gel is a transdermal treatment that will be applied as three single applications to a male subject's arms and shoulders on three different treatment days. The formulation will be a hydro alcoholic gel containing about 1.43% T (14.3 mg T/g gel). About 9 to 14% of the steroid (T or NES) in the gel applied is available to the body. The amount of gel to be applied each application will be approximately 5 mL in volume. The gel application volume will contain 62.5 mg of T that will deliver approximately 6 mg T to the body per day (Swerdloff et al., 2000; Wang et al., 2000). This gel volume will also contain 8.3 mg of NES that will deliver about 0.8 mg of NES to the body per day (NES 8 mg/d + T 60 mg/d (NES8/T60) gel).
  Other Names: NES/T gel; NES8/T60

SUMMARY:
This is a two-center, open-label study conducted in healthy male and female volunteers at two academic research centers. The study will consist of three single applications of the Nestorone (NES) + testosterone (T) combined gel on the shoulders/upper arms of male participants followed 2 hours later by supervised skin contact by the non-dosed female participants on the application site on days 1, 8, and 15. Effect of Washing or Clothing Barrier to the Application will be assessed.

DETAILED DESCRIPTION:
This is a two-center, open-label study conducted in healthy male and female volunteers at two academic research centers. The study will consist of three single applications of the Nestorone (NES) + testosterone (T) combined gel on the shoulders/upper arms of male participants followed 2 hours later by supervised skin contact by the non-dosed female participants on the application site on days 1, 8, and 15.

On day 1, the male participant will wear a 100% cotton T-shirt over the application area before skin contact with the female.

On day 8, the male participant will shower approximately 1 hour and 45 minutes after gel application and engage in skin contact with the female participant (2 hours after gel application) after washing the area with soap and water then drying it. A measurement of residual Nestorone and testosterone will be taken from the male's skin on a single location of the application site using adhesive D-square strips 90 minutes after application (30 minutes before shower/90 minutes after gel application) and 30 minutes after the shower and rubbing (150 minutes after application).

On day 15, there will be no shower or clothing barrier for the male participant before skin contact with the female participant. A measurement of residual Nestorone and testosterone will be taken from a single location of the application using adhesive D-square strips site 90 minutes and 150 minutes after the application.

An end of study/exit visit will occur for both male and female participants two weeks after treatment completion.

ELIGIBILITY:
Inclusion Male participant - Inclusion Criteria

Men who meet all the following criteria will be eligible for enrollment in the trial:

1. Good health as confirmed by medical history, physical examination, and clinical laboratory tests of blood and urine at the time of screening;
2. 18 to 50 years of age;
3. BMI ≥ 18 and < 35 kg/m2;
4. No history of androgen use prior to the first screening visit as follows:

   1. 1 month prior for oral or transdermal androgen,
   2. 3 months prior for Testosterone cypionate or enanthate injection,
   3. 6 months prior for Testosterone undecanoate injection;
5. Agreement to use a recognized effective method of short acting contraception with his partner (i.e. at a minimum use double-barrier method such as a condom with spermicide) during the entire study;
6. In the opinion of the investigator, male subject is willing and able to comply with the protocol;
7. Provision of valid, written and informed consent.

Female participant - Inclusion Criteria

Women who meet all the following criteria will be eligible for enrollment in the trial:

1. Good general health (BMI ≥18 and <30 kg/m2)with no chronic medical conditions that result in periodic exacerbations which require significant medical care;
2. Aged between 18 and 40 years, at the enrollment visit;
3. Not pregnant and not breastfeeding.
4. Agreement to use a recognized effective method of contraception throughout the study
5. Willingness and ability to provide valid, written and informed consent and to comply with the protocol;
6. No desire for pregnancy within the next 6 months.

Exclusion Male participant - Exclusion Criteria

Men who meet any of the following criteria are not eligible for enrollment in the trial:

1. Men participating in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit.
2. Men not living in the catchment area of the study site or within a reasonable travel time from the site.
3. Any clinically significant abnormal findings at screening per the Investigator's medical judgement.
4. Elevated PSA (e.g. levels ≥ 4 ng/mL), according to study site's local laboratory reference normal values for adult men.
5. Abnormal serum chemistry values that may indicate clinically significant liver or kidney dysfunction. Other abnormal laboratory values may also be exclusionary, if so considered by the investigator to be clinically significant.
6. Use of androgens or other anabolic steroids that may affect testosterone measurements
7. Diastolic blood pressure (DBP) ≥ 85 and Systolic blood pressure (SBP) ≥ 135 mm Hg; (BP will be taken three times at approximately 5 minute intervals and the mean of the 3 measurements will be considered).
8. History of hypertension (well-controlled treated hypertension (< 135/85) is allowed).
9. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis.
10. Known hypersensitivity to progestins or testosterone.
11. History of prostate or breast carcinoma
12. Significant lower urinary obstructive symptoms (IPSS > 19).
13. Known history of significant cardiac, renal, hepatic or prostatic disease.
14. History of thromboembolic disease.
15. A serious systemic disease such as diabetes mellitus (including diabetes controlled with treatment), HIV, or morbid obesity.
16. Current active or ongoing Hepatitis infection
17. Known or suspected current alcohol dependence syndrome, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of steroid hormones and study treatment compliance.
18. Known active or chronic dermatitis or other severe skin disorder.
19. Desiring fertility within 6 months of study participation.
20. History of severe depression or other serious mental health disorder.
21. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine will be advised of the relative and temporary hazards that participating in this study may have for their sporting status.

Female participant - Exclusion Criteria

Women who meet any of the following criteria are not eligible for enrollment in the trial:

1. Desire to become pregnant during the study.
2. Breastfeeding
3. Known or suspected current alcoholism or drug abuse.
4. History of thrombosis
5. Serum testosterone outside normal reference ranges by local laboratory standards or evidence of hirsutism (modified Ferriman-Galwey score > 8)
6. Participation in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit.
7. Current pregnancy.
8. Known hypersensitivity to progestins or testosterone.
9. Any clinically significant abnormal findings at screening per the Investigator's medical judgement.
10. Use of androgens or other anabolic steroids that may affect testosterone measurements.
11. Known active or chronic dermatitis or other severe skin disorder.
12. Known or suspected current alcohol dependence syndrome, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of steroid hormones and study treatment compliance.
13. Not living in the catchment area of the study site or within a reasonable travel time from the site.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Bradley Anawalt, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Washington Medical Center & Health Sciences, Seattle, Washington

REFERENCES:
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Bebb RA, Anawalt BD, Christensen RB, Paulsen CA, Bremner WJ, Matsumoto AM. Combined administration of levonorgestrel and testosterone induces more rapid and effective suppression of spermatogenesis than testosterone alone: a promising male contraceptive approach. J Clin Endocrinol Metab. 1996 Feb;81(2):757-62. doi: 10.1210/jcem.81.2.8636300.
- [Background] Brachet C, Vermeulen J, Heinrichs C. Children's virilization and the use of a testosterone gel by their fathers. Eur J Pediatr. 2005 Oct;164(10):646-7. doi: 10.1007/s00431-005-1714-z. Epub 2005 Jul 16. PMID 16025298
- [Background] Brache V, Massai R, Mishell DR, Moo-Young AJ, Alvarez F, Salvatierra AM, Cochon L, Croxatto H, Robbins A, Faundes A. Ovarian function during use of Nestorone(R) subdermal implants. Contraception. 2000 Mar;61(3):199-204. doi: 10.1016/s0010-7824(00)00092-5. PMID 10827334
- [Background] Cummings DE, Bremner WJ. Prospects for new hormonal male contraceptives. Endocrinol Metab Clin North Am. 1994 Dec;23(4):893-922. PMID 7705326
- [Background] de Ronde W, Vogel S, Bui HN, Heijboer AC. Reduction in 24-hour plasma testosterone levels in subjects who showered 15 or 30 minutes after application of testosterone gel. Pharmacotherapy. 2011 Mar;31(3):248-52. doi: 10.1592/phco.31.3.248. PMID 21361734
- [Background] Diaz S, Schiappacasse V, Pavez M, Zepeda A, Moo-Young AJ, Brandeis A, Lahteenmaki P, Croxatto HB. Clinical trial with Nestorone subdermal contraceptive implants. Contraception. 1995 Jan;51(1):33-8. doi: 10.1016/0010-7824(94)00006-i. PMID 7750282
- [Background] Dorman E, Bishai D. Demand for male contraception. Expert Rev Pharmacoecon Outcomes Res. 2012 Oct;12(5):605-13. doi: 10.1586/erp.12.52. PMID 23186401
- [Background] Fraser IS, Weisberg E, Kumar N, Kumar S, Humberstone AJ, McCrossin L, Shaw D, Tsong YY, Sitruk-Ware R. An initial pharmacokinetic study with a Metered Dose Transdermal Systemfor delivery of the progestogen Nestorone as a possible future contraceptive. Contraception. 2007 Dec;76(6):432-8. doi: 10.1016/j.contraception.2007.08.006. Epub 2007 Nov 9. PMID 18061700
- [Background] Handelsman DJ, Conway AJ, Howe CJ, Turner L, Mackey MA. Establishing the minimum effective dose and additive effects of depot progestin in suppression of human spermatogenesis by a testosterone depot. J Clin Endocrinol Metab. 1996 Nov;81(11):4113-21. doi: 10.1210/jcem.81.11.8923869.
- [Background] Haukkamaa M, Laurikka-Routti M, Heikinheimo O, Moo-Young A. Contraception with subdermal implants releasing the progestin ST-1435: a dose-finding study. Contraception. 1992 Jan;45(1):49-55. doi: 10.1016/0010-7824(92)90140-o. PMID 1591921
- [Background] Heinemann K, Saad F, Wiesemes M, White S, Heinemann L. Attitudes toward male fertility control: results of a multinational survey on four continents. Hum Reprod. 2005 Feb;20(2):549-56. doi: 10.1093/humrep/deh574. Epub 2004 Dec 17. PMID 15608042
- [Background] Ilani N, Liu PY, Swerdloff RS, Wang C. Does ethnicity matter in male hormonal contraceptive efficacy? Asian J Androl. 2011 Jul;13(4):579-84. doi: 10.1038/aja.2010.133. Epub 2011 Feb 14. PMID 21317912
- [Background] Ilani N, Roth MY, Amory JK, Swerdloff RS, Dart C, Page ST, Bremner WJ, Sitruk-Ware R, Kumar N, Blithe DL, Wang C. A new combination of testosterone and nestorone transdermal gels for male hormonal contraception. J Clin Endocrinol Metab. 2012 Oct;97(10):3476-86. doi: 10.1210/jc.2012-1384. Epub 2012 Jul 12. PMID 22791756
- [Background] Kamischke A, Ploger D, Venherm S, von Eckardstein S, von Eckardstein A, Nieschlag E. Intramuscular testosterone undecanoate with or without oral levonorgestrel: a randomized placebo-controlled feasibility study for male contraception. Clin Endocrinol (Oxf). 2000 Jul;53(1):43-52. doi: 10.1046/j.1365-2265.2000.01024.x. PMID 10931079
- [Background] Knuth UA, Yeung CH, Nieschlag E. Combination of 19-nortestosterone-hexyloxyphenylpropionate (Anadur) and depot-medroxyprogesterone-acetate (Clinovir) for male contraception. Fertil Steril. 1989 Jun;51(6):1011-8. doi: 10.1016/s0015-0282(16)60735-5. PMID 2524404
- [Background] Kumar N, Koide SS, Tsong Y, Sundaram K. Nestorone: a progestin with a unique pharmacological profile. Steroids. 2000 Oct-Nov;65(10-11):629-36. doi: 10.1016/s0039-128x(00)00119-7. PMID 11108869
- [Background] Kunz GJ, Klein KO, Clemons RD, Gottschalk ME, Jones KL. Virilization of young children after topical androgen use by their parents. Pediatrics. 2004 Jul;114(1):282-4. doi: 10.1542/peds.114.1.282. PMID 15231947
- [Background] Laurikka-Routti M, Haukkamaa M, Heikinheimo O. A contraceptive vaginal ring releasing ethinyl estradiol and the progestin ST-1435: bleeding control, serum steroid concentrations, serum lipids and serum chemistry. Contraception. 1990 Jul;42(1):111-20. doi: 10.1016/0010-7824(90)90095-d. PMID 2387151
- [Background] Mahabadi V, Amory JK, Swerdloff RS, Bremner WJ, Page ST, Sitruk-Ware R, Christensen PD, Kumar N, Tsong YY, Blithe D, Wang C. Combined transdermal testosterone gel and the progestin nestorone suppresses serum gonadotropins in men. J Clin Endocrinol Metab. 2009 Jul;94(7):2313-20. doi: 10.1210/jc.2008-2604. Epub 2009 Apr 14. PMID 19366848
- [Background] Martin CW, Anderson RA, Cheng L, Ho PC, van der Spuy Z, Smith KB, Glasier AF, Everington D, Baird DT. Potential impact of hormonal male contraception: cross-cultural implications for development of novel preparations. Hum Reprod. 2000 Mar;15(3):637-45. doi: 10.1093/humrep/15.3.637. PMID 10686211
- [Background] Merhi ZO, Santoro N. Postmenopausal virilization after spousal use of topical androgens. Fertil Steril. 2007 Apr;87(4):976.e13-5. doi: 10.1016/j.fertnstert.2006.07.1547. Epub 2007 Jan 24. PMID 17254577
- [Background] Miller MG, Rogol AD, Zumbrunnen TL. Secondary exposure to testosterone from patients receiving replacement therapy with transdermal testosterone gels. Curr Med Res Opin. 2012 Feb;28(2):267-9. doi: 10.1185/03007995.2011.652255. Epub 2012 Jan 20. No abstract available. PMID 22185432
- [Background] Nieschlag E, Zitzmann M, Kamischke A. Use of progestins in male contraception. Steroids. 2003 Nov;68(10-13):965-72. doi: 10.1016/s0039-128x(03)00135-1. PMID 14667989
- [Background] Rolf C, Knie U, Lemmnitz G, Nieschlag E. Interpersonal testosterone transfer after topical application of a newly developed testosterone gel preparation. Clin Endocrinol (Oxf). 2002 May;56(5):637-41. doi: 10.1046/j.1365-2265.2002.01529.x. PMID 12030915
- [Background] Shiraishi S, Lee PW, Leung A, Goh VH, Swerdloff RS, Wang C. Simultaneous measurement of serum testosterone and dihydrotestosterone by liquid chromatography-tandem mass spectrometry. Clin Chem. 2008 Nov;54(11):1855-63. doi: 10.1373/clinchem.2008.103846. Epub 2008 Sep 18. PMID 18801940
- [Background] Sitruk-Ware R. Transdermal delivery of steroids. Contraception. 1989 Jan;39(1):1-20. doi: 10.1016/0010-7824(89)90012-7. PMID 2642780
- [Background] Sitruk-Ware R. Transdermal application of steroid hormones for contraception. J Steroid Biochem Mol Biol. 1995 Jun;53(1-6):247-51. doi: 10.1016/0960-0760(95)00055-5. PMID 7626463
- [Background] Sitruk-Ware R, Small M, Kumar N, Tsong YY, Sundaram K, Jackanicz T. Nestorone: clinical applications for contraception and HRT. Steroids. 2003 Nov;68(10-13):907-13. doi: 10.1016/s0039-128x(03)00140-5. PMID 14667982
- [Background] Stahlman J, Britto M, Fitzpatrick S, McWhirter C, Testino SA, Brennan JJ, Zumbrunnen TL. Effect of application site, clothing barrier, and application site washing on testosterone transfer with a 1.62% testosterone gel. Curr Med Res Opin. 2012 Feb;28(2):281-90. doi: 10.1185/03007995.2011.652731. Epub 2012 Jan 25. PMID 22188557
- [Background] Stahlman J, Britto M, Fitzpatrick S, McWhirter C, Testino SA, Brennan JJ, Zumbrunnen TL. Effects of skin washing on systemic absorption of testosterone in hypogonadal males after administration of 1.62% testosterone gel. Curr Med Res Opin. 2012 Feb;28(2):271-9. doi: 10.1185/03007995.2011.652256. Epub 2012 Jan 17. PMID 22185431
- [Background] Stahlman J, Britto M, Fitzpatrick S, McWhirter C, Testino SA, Brennan JJ, Zumbrunnen TL. Serum testosterone levels in non-dosed females after secondary exposure to 1.62% testosterone gel: effects of clothing barrier on testosterone absorption. Curr Med Res Opin. 2012 Feb;28(2):291-301. doi: 10.1185/03007995.2011.652732. Epub 2012 Jan 24. PMID 22188558
- [Background] Swerdloff RS, Wang C, Cunningham G, Dobs A, Iranmanesh A, Matsumoto AM, Snyder PJ, Weber T, Longstreth J, Berman N. Long-term pharmacokinetics of transdermal testosterone gel in hypogonadal men. J Clin Endocrinol Metab. 2000 Dec;85(12):4500-10. doi: 10.1210/jcem.85.12.7045. PMID 11134099
- [Background] Turner L, Conway AJ, Jimenez M, Liu PY, Forbes E, McLachlan RI, Handelsman DJ. Contraceptive efficacy of a depot progestin and androgen combination in men. J Clin Endocrinol Metab. 2003 Oct;88(10):4659-67. doi: 10.1210/jc.2003-030107. PMID 14557437
- [Background] Wallace EM, Wu FC. Effect of depot medroxyprogesterone acetate and testosterone oenanthate on serum lipoproteins in man. Contraception. 1990 Jan;41(1):63-71. doi: 10.1016/0010-7824(90)90127-h. PMID 2137405
- [Background] Wang C, Berman N, Longstreth JA, Chuapoco B, Hull L, Steiner B, Faulkner S, Dudley RE, Swerdloff RS. Pharmacokinetics of transdermal testosterone gel in hypogonadal men: application of gel at one site versus four sites: a General Clinical Research Center Study. J Clin Endocrinol Metab. 2000 Mar;85(3):964-9. doi: 10.1210/jcem.85.3.6437. PMID 10720024
- [Background] Wang C, Wang XH, Nelson AL, Lee KK, Cui YG, Tong JS, Berman N, Lumbreras L, Leung A, Hull L, Desai S, Swerdloff RS. Levonorgestrel implants enhanced the suppression of spermatogenesis by testosterone implants: comparison between Chinese and non-Chinese men. J Clin Endocrinol Metab. 2006 Feb;91(2):460-70. doi: 10.1210/jc.2005-1743. Epub 2005 Nov 8. PMID 16278260
- [Background] Wang C, Shiraishi S, Leung A, Baravarian S, Hull L, Goh V, Lee PW, Swerdloff RS. Validation of a testosterone and dihydrotestosterone liquid chromatography tandem mass spectrometry assay: Interference and comparison with established methods. Steroids. 2008 Dec 12;73(13):1345-52. doi: 10.1016/j.steroids.2008.05.004. Epub 2008 May 21. PMID 18579171
- [Background] Wang C, Swerdloff RS, Iranmanesh A, Dobs A, Snyder PJ, Cunningham G, Matsumoto AM, Weber T, Berman N; Testosterone Gel Study Group. Transdermal testosterone gel improves sexual function, mood, muscle strength, and body composition parameters in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2839-53. doi: 10.1210/jcem.85.8.6747. PMID 10946892
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Background] Wu FC, Balasubramanian R, Mulders TM, Coelingh-Bennink HJ. Oral progestogen combined with testosterone as a potential male contraceptive: additive effects between desogestrel and testosterone enanthate in suppression of spermatogenesis, pituitary-testicular axis, and lipid metabolism. J Clin Endocrinol Metab. 1999 Jan;84(1):112-22. doi: 10.1210/jcem.84.1.5412. PMID 9920070
- [Derived] Yuen F, Wu S, Thirumalai A, Swerdloff RS, Page ST, Liu PY, Dart C, Wu H, Blithe DL, Sitruk-Ware R, Long J, Bai F, Hull L, Bremner WJ, Anawalt BD, Wang C. Preventing secondary exposure to women from men applying a novel nestorone/testosterone contraceptive gel. Andrology. 2019 Mar;7(2):235-243. doi: 10.1111/andr.12577. Epub 2018 Dec 16. PMID 30556332

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 partners were enrolled (13 females and 13 males); Planned enrollment was 24 but study enrolled 26 participants.
Period: Overall Study
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Started | 26
Completed | 24
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The analysis population includes 13 couples - 13 males and 13 females.
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants] — Population: Characteristics were measured for the male subjects and their female partners, and provided separately.
  Participants
    Male Subjects: number analyzed (Participants) | 13
    Male Subjects: <=18 years | 0
    Male Subjects: Between 18 and 65 years | 13
    Male Subjects: >=65 years | 0
    Female Subjects: number analyzed (Participants) | 13
    Female Subjects: <=18 years | 0
    Female Subjects: Between 18 and 65 years | 13
    Female Subjects: >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Characteristics were measured for the male subjects and their female partners, and provided separately.
  years
    Male Subjects: number analyzed (Participants) | 13
    Male Subjects | 29.4 (7.82)
    Female Subjects: number analyzed (Participants) | 13
    Female Subjects | 25.9 (4.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Characteristics were measured for the male subjects and their female partners, and provided separately.
  Participants
    Male Subjects: number analyzed (Participants) | 13
    Male Subjects: Hispanic or Latino | 5
    Male Subjects: Not Hispanic or Latino | 8
    Male Subjects: Unknown or Not Reported | 0
    Female Subjects: number analyzed (Participants) | 13
    Female Subjects: Hispanic or Latino | 6
    Female Subjects: Not Hispanic or Latino | 7
    Female Subjects: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Characteristics were measured for the male subjects and their female partners, and provided separately.
  Participants
    Male Subjects: number analyzed (Participants) | 13
    Male Subjects: American Indian or Alaska Native | 1
    Male Subjects: Asian | 1
    Male Subjects: Native Hawaiian or Other Pacific Islander | 0
    Male Subjects: Black or African American | 3
    Male Subjects: White | 6
    Male Subjects: More than one race | 0
    Male Subjects: Unknown or Not Reported | 2
    Female Subjects: number analyzed (Participants) | 13
    Female Subjects: American Indian or Alaska Native | 0
    Female Subjects: Asian | 1
    Female Subjects: Native Hawaiian or Other Pacific Islander | 0
    Female Subjects: Black or African American | 1
    Female Subjects: White | 7
    Female Subjects: More than one race | 3
    Female Subjects: Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Population: All subjects were enrolled in the United States.
  participants
    United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline (Cavg) for Serum Testosterone Levels in Females After Secondary Exposure to Nestorone + Testosterone Combination Gel
Description: Evaluate in female participants by assessing changes from baseline up to 48 hours for serum testosterone levels in Cavg after secondary exposure to Nestorone + Testosterone Combination Gel summarized for each of the 3 types of skin contact between the man and woman.
Time Frame: Baseline and 48 hours after each intervention (day 1 for t-shirt, day 8 for shower and dried, and day 15 for no shower or t-shirt)
Population: includes female participants that completed the skin contact types
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
ng/dL
  Baseline | 22.84 (8.98)
  With T-shirt Clothing Barrier | 27.12 (9.53)
  Shower and Dried | 29.12 (11.19)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 62.06 (35.68)

2. Secondary Outcome: PK of T in Males After NES/T With a T-shirt and After Washing
Description: PK of testosterone in males after wearing a T shirt and after washing will be compared to serum testosterone PK after application of the combined gel without washing using AUC (0-t, where t is the last time-point with measurable concentration)
Time Frame: Baseline and 24 hours after each intervention (day 1 for t-shirt, day 8 for shower and dried, and day 15 for no shower or t-shirt)
Population: Subjects that had measurements at the respective timepoints were included
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
ng/dL
  With T-shirt Clothing Barrier | 16039.71 (6740.37)
  Shower and Dried | 14297.19 (5539.57)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 15268.13 (5024.31)

3. Secondary Outcome: PK of NES in Males After NES/T With a T-shirt and After Washing
Description: PK of Nestorone in males after wearing a T shirt and after washing will be compared to serum Nestorone PK after application of the combined gel without washing using AUC (0-t, where t is the last time-point with measurable concentration)
Time Frame: as for outcome 2
Population: Subjects that had measurements at the respective timepoints were included
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
pg/dL
  With T-shirt Clothing Barrier | 5376.41 (6730.65)
  Shower and Dried | 1913.47 (2178.22)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 4550.17 (4448.20)

4. Secondary Outcome: Average Testosterone Levels 90 and 150 Minutes After Each Application in Men
Description: Average testosterone levels 90 and 150 minutes after each application in men (over a 15 day period) as measured by adhesive D-square strips with showering (Visit 5) and without showering (Visit 7).
Time Frame: Visits 5 and 7 (Days 8 and 15)
Population: Subjects that had measurements at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: T (microg)
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
T (microg)
  Visit 5, 90 min (With Shower) | 17.39 (8.85)
  Visit 5, 150 min (With Shower) | 0.24 (0.44)
  Visit 7, 90 min (Without Shower): number analyzed (Participants) | 12
  Visit 7, 90 min (Without Shower) | 17.69 (13.58)
  Visit 7, 150 min (Without Shower): number analyzed (Participants) | 12
  Visit 7, 150 min (Without Shower) | 8.23 (7.10)

5. Secondary Outcome: Average Nestorone Levels 90 and 150 Minutes After Each Application in Men
Description: Average Nestorone levels 90 and 150 minutes after each application in men (over a 15 day period) as measured by adhesive D-square strips with showering (Visit 5) and without showering (Visit 7).
Time Frame: Visits 5 and 7 (Days 8 and 15)
Population: Subjects that had measurements at the respective timepoints were analyzed
Measure: Mean (Standard Deviation); unit: NES (microg)
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
NES (microg)
  Visit 5, 90 min (With Shower) | 2.19 (1.30)
  Visit 5, 150 min (With Shower) | 0.04 (0.08)
  Visit 7, 90 min (Without Shower): number analyzed (Participants) | 12
  Visit 7, 90 min (Without Shower) | 1.98 (1.52)
  Visit 7, 150 min (Without Shower): number analyzed (Participants) | 12
  Visit 7, 150 min (Without Shower) | 1.03 (0.99)

6. Secondary Outcome: Incidence of Adverse Events and Serious Adverse Events for Males
Description: Male AEs
Time Frame: 31 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
Participants | 1

7. Secondary Outcome: Incidence of Adverse Events and Serious Adverse Events for Females
Description: Female AEs
Time Frame: 31 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
Participants | 5

8. Secondary Outcome: Changes From Baseline in Hematology Safety Labs for Females
Description: Changes from baseline in hematology parameters for females measured at Screening (Day -28 to 0) and Visit 7 (Day 15)
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least on post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
10^3 cells/uL
  Basophils: number analyzed (Participants) | 9
  Basophils | -0.007 (0.0173)
  Eosinophils: number analyzed (Participants) | 9
  Eosinophils | 0.026 (0.0400)
  Lymphocytes: number analyzed (Participants) | 9
  Lymphocytes | -0.216 (0.7371)
  Monocytes: number analyzed (Participants) | 9
  Monocytes | 0.024 (0.0872)
  Neutrophils: number analyzed (Participants) | 9
  Neutrophils | -1.321 (1.0245)
  Platelet Count: number analyzed (Participants) | 11
  Platelet Count | -3.2 (28.75)
  White Blood Cells: number analyzed (Participants) | 12
  White Blood Cells | -1.083 (1.4826)

9. Primary Outcome: Changes From Baseline (Cmin) for Serum Testosterone Levels in Females After Secondary Exposure to Nestorone + Testosterone Combination Gel
Description: Evaluate in female participants by assessing changes from baseline up to 48 hours for serum testosterone levels in Cmin after secondary exposure to Nestorone + Testosterone Combination Gel summarized for each of the 3 types of skin contact between the man and woman.
Time Frame: as for outcome 1
Population: includes female participants that completed the skin contact types
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
ng/dL
  Baseline | 20.63 (9.13)
  With T-shirt Clothing Barrier | 21.26 (9.04)
  Shower and Dried | 23.27 (10.88)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 22.94 (10.07)

10. Primary Outcome: Changes From Baseline (Cmax) for Serum Testosterone Levels in Females After Secondary Exposure to Nestorone + Testosterone Combination Gel
Description: Evaluate in female participants by assessing changes from baseline up to 48 hours for serum testosterone levels in Cmax after secondary exposure to Nestorone + Testosterone Combination Gel summarized for each of the 3 types of skin contact between the man and woman.
Time Frame: as for outcome 1
Population: includes female participants that completed the skin contact types
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
ng/dL
  Baseline | 31.8 (12.0)
  With T-shirt Clothing Barrier | 39.4 (12.9)
  Shower and Dried | 48.1 (23.5)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 123.0 (85.3)

11. Primary Outcome: Changes From Baseline (Cmin) for Serum Nestorone Levels in Females After Secondary Exposure to Nestorone + Testosterone Combination Gel
Description: Evaluate in female participants by assessing changes from baseline up to 48 hours for serum Nestorone levels in Cmin after secondary exposure to Nestorone + Testosterone Combination Gel summarized for each of the 3 types of skin contact between the man and woman.
Time Frame: as for outcome 1
Population: includes female participants that had measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
pg/dL
  Baseline: number analyzed (Participants) | 12
  Baseline | 0 (0)
  With T-shirt Clothing Barrier | 0 (0)
  Shower and Dried | 0 (0)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 0 (0)

12. Primary Outcome: Changes From Baseline (Cmax) for Serum Nestorone Levels in Females After Secondary Exposure to Nestorone + Testosterone Combination Gel
Description: Evaluate in female participants by assessing changes from baseline up to 48 hours for serum Nestorone levels in Cmax after secondary exposure to Nestorone + Testosterone Combination Gel summarized for each of the 3 types of skin contact between the man and woman.
Time Frame: as for outcome 1
Population: includes female participants that had measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
pg/dL
  Baseline: number analyzed (Participants) | 12
  Baseline | 0 (0)
  With T-shirt Clothing Barrier | 4.19 (15.10)
  Shower and Dried | 3.60 (10.07)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 29.3 (35.5)

13. Primary Outcome: Changes From Baseline (Cavg) for Serum Nestorone Levels in Females After Secondary Exposure to Nestorone + Testosterone Combination Gel
Description: Evaluate in female participants by assessing changes from baseline up to 48 hours for serum Nestorone levels in Cavg after secondary exposure to Nestorone + Testosterone Combination Gel summarized for each of the 3 types of skin contact between the man and woman.
Time Frame: as for outcome 1
Population: includes female participants that had measurements at the specified timepoints
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
pg/dL
  Baseline: number analyzed (Participants) | 12
  Baseline | 0 (0)
  With T-shirt Clothing Barrier | 0.97 (3.51)
  Shower and Dried | 0.47 (1.51)
  No Intervention: number analyzed (Participants) | 12
  No Intervention | 8.12 (10.91)

14. Secondary Outcome: Changes From Baseline in Hematology Safety Labs for Males
Description: Changes from baseline in hematology parameters for males measured at Screening (Day -28 to 0) and Visit 7 (Day 15)
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
10^3 cells/uL
  Basophils: number analyzed (Participants) | 9
  Basophils | 0.000 (0.0150)
  Eosinophils: number analyzed (Participants) | 9
  Eosinophils | -0.002 (0.0286)
  Lymphocytes: number analyzed (Participants) | 9
  Lymphocytes | 0.416 (0.6456)
  Monocytes: number analyzed (Participants) | 9
  Monocytes | -0.077 (0.5130)
  Neutrophils: number analyzed (Participants) | 9
  Neutrophils | 0.239 (0.5169)
  Platelet Count: number analyzed (Participants) | 12
  Platelet Count | 0.7 (41.15)
  White Blood Cells: number analyzed (Participants) | 12
  White Blood Cells | 0.026 (1.4054)

15. Secondary Outcome: Changes From Baseline in Hematology Safety Labs for Females
Description: Changes from baseline in hematology parameters for females measured at Screening (Day -28 to 0) and Visit 7 (Day 15)
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
g/L
  Ery. Mean Corpuscular HGB Concentration: number analyzed (Participants) | 12
  Ery. Mean Corpuscular HGB Concentration | -2.9 (8.32)
  Hemoglobin: number analyzed (Participants) | 12
  Hemoglobin | -12.8 (6.97)

16. Secondary Outcome: Changes From Baseline in Hematology Safety Labs for Males
Description: Changes from baseline in hematology parameters for males measured at Screening (Day -28 to 0) and Visit 7 (Day 15)
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
g/L
  Ery. Mean Corpuscular HGB Concentration: number analyzed (Participants) | 12
  Ery. Mean Corpuscular HGB Concentration | 0.4 (7.48)
  Hemoglobin: number analyzed (Participants) | 12
  Hemoglobin | -8.8 (7.89)

17. Secondary Outcome: Changes From Baseline in Clinical Chemistry Safety Labs for Females
Description: Changes from baseline in clinical chemistry parameters for females measured at Screening (Day -28 to 0) and Visit 7 (Day 15)
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
U/L
  ALT/SGPT: number analyzed (Participants) | 12
  ALT/SGPT | -1.8 (3.55)
  AST/SGOT: number analyzed (Participants) | 12
  AST/SGOT | -1.3 (2.74)
  Alkaline Phosphatase: number analyzed (Participants) | 12
  Alkaline Phosphatase | -3.9 (6.22)

18. Secondary Outcome: Changes From Baseline in Clinical Chemistry Safety Labs for Males
Description: Changes from baseline in clinical chemistry parameters for males measured at Screening (Day -28 to 0) and Visit 7 (Day 15)
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
U/L
  ALT/SGPT: number analyzed (Participants) | 12
  ALT/SGPT | -1.9 (5.81)
  AST/SGOT: number analyzed (Participants) | 12
  AST/SGOT | -4.0 (4.05)
  Alkaline Phosphatase: number analyzed (Participants) | 12
  Alkaline Phosphatase | -10.4 (11.43)

19. Secondary Outcome: Changes From Baseline in Clinical Chemistry Safety Labs for Females
Description: as for outcome 17
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
g/L
  Albumin: number analyzed (Participants) | 12
  Albumin | -3.1 (2.19)
  Total Protein: number analyzed (Participants) | 12
  Total Protein | -4.9 (3.55)

20. Secondary Outcome: Changes From Baseline in Clinical Chemistry Safety Labs for Males
Description: as for outcome 18
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
g/L
  Albumin: number analyzed (Participants) | 12
  Albumin | -5.2 (3.74)
  Total Protein: number analyzed (Participants) | 12
  Total Protein | -7.5 (6.45)

21. Secondary Outcome: Changes From Baseline in Clinical Chemistry Safety Labs for Females
Description: as for outcome 17
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
mmol/L
  BUN: number analyzed (Participants) | 12
  BUN | 0.060 (0.8199)
  Bicarbonate: number analyzed (Participants) | 12
  Bicarbonate | -1.2 (2.37)
  Calcium: number analyzed (Participants) | 12
  Calcium | -0.064 (0.0720)
  Chloride: number analyzed (Participants) | 12
  Chloride | 1.8 (1.66)
  Glucose: number analyzed (Participants) | 12
  Glucose | 0.375 (0.5547)
  Potassium: number analyzed (Participants) | 12
  Potassium | -0.02 (0.292)
  Sodium: number analyzed (Participants) | 12
  Sodium | -0.6 (2.23)

22. Secondary Outcome: Changes From Baseline in Clinical Chemistry Safety Labs for Males
Description: as for outcome 18
Time Frame: Screening and Visit 7, up to 43 days
Population: only includes subjects who had both baseline and at least one post-baseline non-missing data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
mmol/L
  BUN: number analyzed (Participants) | 12
  BUN | -0.713 (1.4980)
  Bicarbonate: number analyzed (Participants) | 12
  Bicarbonate | -1.9 (3.26)
  Calcium: number analyzed (Participants) | 12
  Calcium | -0.141 (0.1554)
  Chloride: number analyzed (Participants) | 12
  Chloride | 3.3 (3.39)
  Glucose: number analyzed (Participants) | 12
  Glucose | 0.614 (1.1085)
  Potassium: number analyzed (Participants) | 12
  Potassium | -0.33 (0.308)
  Sodium: number analyzed (Participants) | 12
  Sodium | 0.2 (2.44)

23. Secondary Outcome: Percentage of Females With Increased (Relative to Baseline) Hirsutism at Each Visit.
Description: Female hirsutism changes assessed at Screening, Visits 4, 6, 8, and 9
Time Frame: Screening, Visit 4 (Day 3), Visit 6 (Day 10), Visit 8 (Day 17), and Visit 9 (Day 31)
Population: females that were assessed are included
Measure: Count of Participants; unit: Participants
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
Participants
  # of Subjects with increase at Visit 4: number analyzed (Participants) | 12
  # of Subjects with increase at Visit 4 | 0
  # of Subjects with increase at Visit 6 | 0
  # of Subjects with increase at Visit 8: number analyzed (Participants) | 11
  # of Subjects with increase at Visit 8 | 0
  # of Subjects with increase at Visit 9: number analyzed (Participants) | 12
  # of Subjects with increase at Visit 9 | 0

24. Secondary Outcome: Percentage of Females With Increased (Relative to Baseline) Acne at Each Visit.
Description: Female acne changes assessed at Screening, Visits 4, 6, 8, and 9
Time Frame: Screening, Visit 4 (Day 3), Visit 6 (Day 10), Visit 8 (Day 17), and Visit 9 (Day 31)
Population: subjects that had assessments completed at the respective visits were included
Measure: Count of Participants; unit: Participants
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel
Number analyzed (Participants) | 13
Participants
  # of Subjects with increased Facial Acne at Visit 4: number analyzed (Participants) | 12
  # of Subjects with increased Facial Acne at Visit 4 | 0
  # of Subjects with increased Facial Acne at Visit 6 | 1
  # of Subjects with increased Facial Acne at Visit 8: number analyzed (Participants) | 12
  # of Subjects with increased Facial Acne at Visit 8 | 1
  # of Subjects with increased Facial Acne at Visit 9 | 0
  # of Subjects with increased Back Acne at Visit 4: number analyzed (Participants) | 12
  # of Subjects with increased Back Acne at Visit 4 | 0
  Subjects with increased Back Acne at Visit 6 | 1
  Subjects with increased Back Acne at Visit 8: number analyzed (Participants) | 12
  Subjects with increased Back Acne at Visit 8 | 1
  Subjects with increased Back Acne at Visit 9 | 2
  Subjects with increased Chest Acne at Visit 4: number analyzed (Participants) | 12
  Subjects with increased Chest Acne at Visit 4 | 0
  Subjects with increased Chest Acne at Visit 6 | 0
  Subjects with increased Chest Acne at Visit 8: number analyzed (Participants) | 12
  Subjects with increased Chest Acne at Visit 8 | 0
  Subjects with increased Chest Acne at Visit 9 | 0

ADVERSE EVENTS:
Time Frame: 5 months
Description: No change from clinicaltrials.gov definition.
Groups:
- Male Subjects: Includes male participants only.
- Female Subjects: Includes female partners of the male participants.
Arm/Group | Nestorone (NES) + Testosterone (T) Combined Gel | Male Subjects | Female Subjects
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/26 | 1/13 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nestorone (NES) + Testosterone (T) Combined Gel (N=26) | Male Subjects (N=13) | Female Subjects (N=13)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 2 (3)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT02994602/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT02994602/SAP_001.pdf